CLINICAL TRIAL: NCT04798014
Title: Home-Reported Outcomes in People With Cystic Fibrosis (CF) Taking Highly Effective Cystic Fibrosis Transmembrane Conductance Regulator (CFTR) Modulator Therapy
Brief Title: HERO-2: Home-Reported Outcomes With CFTR Modulator Therapy
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Folia Health (Industry); Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Cynthia Brown, Professor of Clinical Medicine, Indiana University
Other Study IDs: 11375
Record Dates: First submitted 2021-03-11; First posted 2021-03-15 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Cystic Fibrosis
Keywords: Trikafta; Triple Combination Therapy; Folia Health
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational cohort study, using data from Folia Health and the Cystic Fibrosis Foundation Patient Registry (CFFPR). Individuals taking elexacaftor/tezacaftor/ivacaftor (ETI) may be enrolled through the Folia application. During the 12-month study period, participants will be asked to track their routine treatment and medication usage, daily symptoms, and monthly review with validated patient-reported outcome (PRO) questionnaires. Participants will also be asked to self-report instances of changes to their treatment plan, and pulmonary exacerbations. There are no study-associated site visits.

DETAILED DESCRIPTION:
This study will be a prospective, observational cohort study to investigate the changes in lung function among individuals who have made treatment changes after initiating treatment with elexacaftor/tezacaftor/ivacaftor (ETI). Data will be collected from Folia Health, and the Cystic Fibrosis Foundation Patient Registry (CFFPR) for participants who are registered. Participation in the study will occur through the Folia application where study participants will be directed to a specific HERO-2 study dashboard. Individuals (n=860) taking ETI may be enrolled at participating sites, through social media recruitment or from existing users of Folia Health. During the 12-month study period, participants will be asked to track their routine treatment and medication usage, daily symptoms, and monthly review with validated CF patient-reported outcome (PRO) questionnaires. Participants will also be asked to self-report instances of changes to their treatment plan, and pulmonary exacerbations. Data collected within Folia will be linked to the CFFPR for individual outcomes with regards to clinical data including anthropometric measures, lung function, complications, and IV-treated pulmonary exacerbations. This study will not provide or recommend any treatment recommendations. All direction for medication usage is solely at the discretion of the patient's physician in accordance with their usual practice.

The primary objective for the study will be to evaluate changes in lung function as measured by forced expiratory volume over one second (FEV1) percent predicted in individuals who report making at least one change to chronic daily respiratory therapies upon study entry and during the 12 month follow up compared to those who do not make changes to chronic daily therapies. Secondary endpoints will include a measurement of the proportion of individuals making changes to chronic daily therapy, the need to resume chronic daily therapy, health-related quality of life, symptom severity and symptom frequency, and pulmonary exacerbations requiring IV antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (and assent when applicable) obtained from subject or subject's legal guardian.
* Is willing and able to adhere to protocol requirements.
* ≥ 12 years of age at enrollment.
* Diagnosed with CF.
* Prescribed ETI for an on-label indication.
* Participant has access to a mobile phone or tablet (iPhone or Android platform) or computer.
* Participant has access to an internet connection.

Exclusion Criteria:

* Participant is enrolled in the randomized portion of the SIMPLIFY study (NCT04378153).
* Participant does not have access to the necessary technology.
* Participant is a recipient of a solid organ transplant (i.e. lung, liver, pancreas, kidney).
* Participant cannot communicate in English.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals diagnosed with Cystic Fibrosis, and who are on ETI through an FDA-labeled indication are eligible for this study. Study participants will be using Folia Health, a web-based application to track daily care and must have access to a mobile phone or computer with an internet connection.
Sampling Method: Non-Probability Sample
Enrollment: 860 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Change in FEV1 percent predicted | 12 months
  The primary outcome measure of this study is change in FEV1 percent predicted at 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States